CLINICAL TRIAL: NCT05459558
Title: A Randomized, Controlled, Single-Blind Clinical Study to Investigate the Tooth Stain Removal Efficacy of Two Experimental Potassium Nitrate Dentifrices in Subjects With Extrinsic Dental Stain Compared to a Standard Dentifrice Control When Used Twice Daily for 8 Weeks
Brief Title: Clinical Study to Investigate the Tooth Stain Removal Efficacy of Two Experimental Toothpastes Compared to a Standard Toothpaste When Used Twice Daily for 8 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300024
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Dentifrice 1 (Experimental): Randomized participants will brush their teeth with the experimental dentifrice (covering the entire length of the toothbrush), twice daily (morning and evening) for 2 minutes for 8 weeks.
  Interventions: Drug: Experimental Dentifrice 1
- Experimental Dentifrice 2 (Experimental): Randomized participants will brush their teeth with the experimental dentifrice (covering the entire length of the toothbrush), twice daily (morning and evening) for 2 minutes for 8 weeks.
  Interventions: Drug: Experimental Dentifrice 2
- Reference Dentifrice (Active Comparator): Randomized participants will brush their teeth with the Reference dentifrice (covering the entire length of the toothbrush), twice daily (morning and evening) for 2 minutes for 8 weeks.
  Interventions: Drug: Reference Dentifrice

INTERVENTIONS:
Drug: Experimental Dentifrice 1 — 5 percent (%) potassium nitrate (KNO3) dentifrice with 1% alumina and 5% sodium tripolyphosphate (STP).
  Arms: Experimental Dentifrice 1
Drug: Experimental Dentifrice 2 — 5% KNO3 dentifrice with 1% alumina, 5% STP and 2% high cleaning silica.
  Arms: Experimental Dentifrice 2
Drug: Reference Dentifrice — Regular Fluoride Dentifrice.
  Arms: Reference Dentifrice

SUMMARY:
The aim of this study is to investigate the stain removal efficacy of 2 experimental anti-dentin hypersensitivity (DH) dentifrices with four and eight weeks twice daily use. A daily use, regular fluoride dentifrice will be included as a reference dentifrice.

DETAILED DESCRIPTION:
This will be a single-center, 8-week, randomized, controlled, single-blind, three treatment-arm, parallel design, stratified clinical study in healthy volunteers with a propensity to form dental stain. It has been designed to investigate changes in tooth stain and color, following twice-daily use of two experimental dentifrices, after four and eight weeks twice daily use; a regular fluoride dentifrice will be included as reference dentifrice. Sufficient participants will be screened to randomize approximately 300 participants to study treatment to ensure approximately 270 participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, product usage requirements, study procedures and lifestyle restrictions.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history (for example, a medical condition confirmed to be causing xerostomia),or upon oral examination, that would impact the participant's safety, wellbeing or the outcomes of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Participant with generally good oral health with:

  1. At least 16 natural (vital) teeth including 11 of the 12 anterior teeth.
  2. Facial surfaces of all anterior teeth (maxillary and mandibular) and lingual surfaces of anterior teeth (mandibular only) gradable for MLSI with no significant calculus or large restorations as judged by the clinical examiner.
  3. Presence of extrinsic dental stain (formed on the surface of the teeth) as determined from a gross visual examination which, in the opinion of the clinical examiner, originates from the diet and/or use of tobacco products.
  4. Facial surfaces of central and lateral maxillary incisors gradable for tooth shade (free of cervical margin defects and restorations which could impact assessment), as judged by the clinical examiner.
  5. Baseline Total MLSI (Area x Intensity) greater than or equal to (>=)15 for the facial surfaces of the 12 anterior teeth.
  6. Baseline mean tooth shade (VITA Bleachedguide 3D-MASTER) >=11 on the facial surfaces of the 4 maxillary incisors.

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of study entry and/or during study participation or who has previously been enrolled in this study.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant who is pregnant (self-reported) or intending to become pregnant during the study.
* Participant who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
* Participant who is unwilling or, in the opinion of the investigator or medically qualified designee, unable to comply with the requirements and/or lifestyle restrictions of the study.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant with Oral Soft Tissue (OST) examination findings at Screening which, in the opinion of the investigator, could interfere with the conduct of the study (for example, stomatitis, open sores, lesions, cavitied caries lesions, redness or swelling.
* Participant using daily oral care products and/or taking daily doses of medications/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with study outcomes, specifically:

  1. currently daily use of mouthwashes containing ingredients known to cause tooth stain (for example, chlorhexidine or cetylpyridinium chloride),
  2. past or current use of minocycline,
  3. use of tetracycline or doxycycline within 30 days of screening and/or during the study,
  4. medications known to cause tooth stain (for example, drugs or supplements containing metal ions known to increase enamel staining).
* Participant who has used any professionally-dispensed tooth whitening products 6 months prior to baseline or any over-the-counter products (including peroxide- or covarine blue-containing dentifrice, but not other daily use whitening dentifrices) 3 months prior to baseline.
* Specific exclusions for assessment teeth:

  1. Non-vital tooth.
  2. Tooth with evidence of current or recent carious lesions.
  3. Tooth used as an abutment for fixed or partial dentures.
  4. Tooth adjacent to fixed retainers and fixed or removable orthodontic appliances.
  5. Tooth with surface irregularities, cracked enamel, discoloration due to trauma or orthodontic treatment, tetracycline stain, restorations or hyper-/hypoplastic areas, which, in the opinion of the clinical examiner, grading of extrinsic dental stain and tooth shade.
  6. Tooth with a crown or veneer.
  7. Tooth with exposed dentine which, in the opinion of the investigator, could impact grading of extrinsic dental stain and tooth shade.
* General oral exclusions:

  1. Generalized severe gingivitis or advanced periodontal disease; treatment of periodontal disease (including surgery) within 12 months of screening; scaling or root planning within 3 months of screening.
  2. Any oral condition requiring immediate care.
  3. Having received a dental prophylaxis within 8 weeks of screening.
* Participant who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research Center (c/o Family & Cosmetic Dentistry), Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be grant-ed, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in the United States of America.
Pre-assignment Details: A total of 281 participants were screened, 280 participants were enrolled, and 279 participants were randomized to a treatment (93 participants in Experimental Dentifrice 1, 92 participants in Experimental Dentifrice 2, and 94 participants in the Reference Dentifrice groups). A total of 272 randomized participants completed the study.
Groups:
- Experimental Dentifrice 1: Randomized participants were instructed to brush their teeth with the experimental dentifrice 1 (5 percent [%] potassium nitrate [KNO3] dentifrice with 1% alumina and 5% sodium tripolyphosphate [STP]), twice daily (morning and evening) for 2 minutes for 8 weeks.
- Experimental Dentifrice 2: Randomized participants were instructed to brush their teeth with the experimental dentifrice 2 (5% KNO3 dentifrice with 1% alumina, 5% STP and 2% high cleaning silica), twice daily (morning and evening) for 2 minutes for 8 weeks.
- Reference Dentifrice: Randomized participants were instructed to brush their teeth with the reference dentifrice (Regular Fluoride Dentifrice), twice daily (morning and evening) for 2 minutes for 8 weeks.
Period: Overall Study
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Started | 93 | 92 | 94
Completed | 92 | 91 | 89
Not Completed | 1 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Scheduling issue | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one post baseline efficacy assessment.
Groups:
- Experimental Dentifrice 1: Randomized participants were instructed to brush their teeth with the experimental dentifrice 1 (5% KNO3 dentifrice with 1% alumina and 5% STP), twice daily (morning and evening) for 2 minutes for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice | Total
Number analyzed (Participants) | 92 | 91 | 90 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.92) | 39.5 (13.73) | 40.5 (13.98) | 41.2 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 59 | 161
  Male | 40 | 41 | 31 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 10 | 27
  Not Hispanic or Latino | 82 | 84 | 80 | 246
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 7 | 5 | 6 | 18
  Asian - Central/South Asian Heritage | 2 | 1 | 3 | 6
  Asian - East Asian Heritage | 1 | 1 | 1 | 3
  White - Arabic/North African Heritage | 1 | 1 | 1 | 3
  White - White/Caucasian/European Heritage | 81 | 83 | 79 | 243

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Total Modified Lobene Stain Index (MLSI) Score at Week 8
Description: Extrinsic dental stain area and its intensity were assessed on the facial surfaces of the 6 maxillary and 6 mandibular anterior teeth and the lingual surfaces of the 6 mandibular anterior teeth. MLSI score= Area score multiplied by Intensity score. Area and intensity of extrinsic dental stain were scored separately for each tooth on the scale 0 to 3, where 0= area with no stain, 1= Stain covering up to one third of area and light intensity stain, 2= Stain covering up to two thirds of area and moderate intensity stain, 3= Stain covering more than two thirds of area and heavy intensity stain. MLSI score ranged from 0 to 9. Mean Total MLSI Score = Mean of MLSI score across all evaluable tooth surfaces for the participant with a range from 0 to 9, where a lower score indicated an improvement. Change from Baseline was calculated by subtracting the Baseline value from the Week 8 value.
Time Frame: Baseline and Week 8
Population: mITT Population. Only those participants available at the indicated timepoint were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | -2.33 (0.048) | -2.42 (0.049) | -0.38 (0.049)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1; Test for non-zero within group change from Baseline; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach
Statistical Analysis 2: Comparison: Experimental Dentifrice 2; Test for non-zero within group change from Baseline; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach

2. Secondary Outcome: Change From Baseline in Mean Total MLSI Score at Week 4
Description: Extrinsic dental stain area and its intensity were assessed on the facial surfaces of the 6 maxillary and 6 mandibular anterior teeth and the lingual surfaces of the 6 mandibular anterior teeth. MLSI score = Area score multiplied by Intensity score. Area and intensity of extrinsic dental stain were scored separately for each tooth on the scale 0 to 3, where 0= area with no stain, 1= Stain covering up to one third of area and light intensity stain, 2= Stain covering up to two thirds of area and moderate intensity stain, 3= Stain covering more than two thirds of area and heavy intensity stain. MLSI score ranged from 0 to 9. Mean Total MLSI Score = Mean of MLSI score across all evaluable tooth surfaces for the participant with a range from 0 to 9, where a lower score indicated an improvement. Change from Baseline was calculated by subtracting the Baseline value from the Week 4 value.
Time Frame: Baseline and Week 4
Population: mITT Population.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 90
score on a scale | -1.94 (0.046) | -1.93 (0.046) | -0.19 (0.047)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1; Test for non-zero within group change from Baseline; Test type: Superiority; p < 0.0001, Mixed Models with Repeated Measures
Statistical Analysis 2: Comparison: Experimental Dentifrice 2; Test for non-zero within group change from Baseline; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

3. Secondary Outcome: Change From Baseline in Mean Total MLSI Score at Weeks 4 and 8
Description: Extrinsic dental stain area and its intensity were assessed on the facial surfaces of the 6 maxillary and 6 mandibular anterior teeth and the lingual surfaces of the 6 mandibular anterior teeth. MLSI score = Area score multiplied by Intensity score. Area and intensity of extrinsic dental stain were scored separately for each tooth on the scale 0 to 3, where 0= area with no stain, 1= Stain covering up to one third of area and light intensity stain, 2= Stain covering up to two thirds of area and moderate intensity stain, 3= Stain covering more than two thirds of area and heavy intensity stain. MLSI score ranged from 0 to 9. Mean Total MLSI Score = Mean of MLSI score across all evaluable tooth surfaces for the participant with a range from 0 to 9, where a lower score indicated an improvement. Change from Baseline was calculated by subtracting the Baseline value from the value at indicated timepoints.
Time Frame: Baseline, Week 4 and Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 90
score on a scale
  Week 4 | -1.94 (0.046) | -1.93 (0.046) | -0.19 (0.047)
  Week 8: number analyzed (Participants) | 92 | 91 | 89
  Week 8 | -2.33 (0.048) | -2.42 (0.049) | -0.38 (0.049)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-1.88 to -1.62], Standard Error of Mean 0.066
Statistical Analysis 2: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-1.87 to -1.61], Standard Error of Mean 0.066
Statistical Analysis 3: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-2.08 to -1.81], Standard Error of Mean 0.069
Statistical Analysis 4: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-2.18 to -1.90], Standard Error of Mean 0.069

4. Secondary Outcome: Change From Baseline in Mean VITA Shade Score (Examiner Assessed) at Weeks 4 and 8
Description: Tooth shade (color) of the facial surfaces of the four central and lateral maxillary incisors was assessed by a trained clinical examiner using the VITA Bleached guide 3D-MASTER. It used a value-ranked ordered scale from 1 (the lightest) to 29 (the darkest). The shade level of each tooth surface was scored visually by the clinical examiner with reference to the Bleached guide, where lower score indicated improvement. Change from Baseline was calculated by subtracting the Baseline value from the value at indicated timepoints.
Time Frame: Baseline, Week 4 and Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 90
score on a scale
  Week 4 | -0.81 (0.068) | -0.59 (0.068) | 0.01 (0.069)
  Week 8: number analyzed (Participants) | 92 | 91 | 89
  Week 8 | -1.73 (0.134) | -1.85 (0.134) | -0.04 (0.136)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.00 to -0.62], Standard Error of Mean 0.097
Statistical Analysis 2: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.79 to -0.41], Standard Error of Mean 0.097
Statistical Analysis 3: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-2.06 to -1.31], Standard Error of Mean 0.190
Statistical Analysis 4: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — p-value adjusted for multiplicity using Graphical Approach; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-2.19 to -1.44], Standard Error of Mean 0.191

5. Secondary Outcome: Change From Baseline in Mean Total MLSI Score in Gingival Sites, Interproximal Sites and Body Sites at Weeks 4 and 8
Description: Extrinsic dental stain area and its intensity were assessed at the specific tooth sites (Gingival site: Crescent-shaped band, adjacent to the free margin of the gingiva and extending to the crest of the interdental papillae of the adjacent teeth. Body Site: The remainder of the tooth surface). MLSI score= Area score multiplied by Intensity score. Area and intensity of extrinsic dental stain was scored separately for each tooth on the scale 0 to 3, where 0= area with no stain, 1= Stain covering up to one third area and light intensity stain, 2= Stain covering up to two thirds area and moderate intensity stain, 3= Stain covering more than two thirds area and heavy intensity stain. MLSI score ranged from 0 to 9. Mean Total MLSI Score= Mean of MLSI score across all evaluable tooth surfaces for the participant with a range from 0 to 9, where a lower score indicated an improvement. Change from Baseline was calculated by subtracting the Baseline value from the value at indicated timepoints.
Time Frame: Baseline, Week 4 and Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 90
score on a scale
  Gingival Sites, Week 4 | -2.39 (0.064) | -2.40 (0.065) | -0.17 (0.065)
  Gingival Sites, Week 8: number analyzed (Participants) | 92 | 91 | 89
  Gingival Sites, Week 8 | -2.96 (0.067) | -3.09 (0.067) | -0.46 (0.068)
  Interproximal Sites, Week 4 | -2.27 (0.055) | -2.25 (0.056) | -0.20 (0.056)
  Interproximal Sites, Week 8: number analyzed (Participants) | 92 | 91 | 89
  Interproximal Sites, Week 8 | -2.69 (0.057) | -2.81 (0.057) | -0.40 (0.058)
  Body Sites, Week 4 | -0.82 (0.046) | -0.84 (0.047) | -0.20 (0.047)
  Body Sites, Week 8: number analyzed (Participants) | 92 | 91 | 89
  Body Sites, Week 8 | -0.95 (0.043) | -0.96 (0.043) | -0.26 (0.043)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Gingival Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-2.41 to -2.05], Standard Error of Mean 0.092
Statistical Analysis 2: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Gingival Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-2.41 to -2.05], Standard Error of Mean 0.092
Statistical Analysis 3: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Gingival Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-2.69 to -2.31], Standard Error of Mean 0.095
Statistical Analysis 4: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Gingival Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-2.81 to -2.44], Standard Error of Mean 0.095
Statistical Analysis 5: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Interproximal Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-2.22 to -1.91], Standard Error of Mean 0.079
Statistical Analysis 6: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Interproximal Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-2.20 to -1.89], Standard Error of Mean 0.079
Statistical Analysis 7: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Interproximal Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-2.45 to -2.13], Standard Error of Mean 0.081
Statistical Analysis 8: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Interproximal Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-2.57 to -2.25], Standard Error of Mean 0.082
Statistical Analysis 9: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Body Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.76 to -0.50], Standard Error of Mean 0.066
Statistical Analysis 10: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Body Sites, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.77 to -0.51], Standard Error of Mean 0.066
Statistical Analysis 11: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Body Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.81 to -0.57], Standard Error of Mean 0.061
Statistical Analysis 12: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Body Sites, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.81 to -0.57], Standard Error of Mean 0.061

6. Secondary Outcome: Change From Baseline in Mean MLSI (Area) and MLSI (Intensity) at Weeks 4 and 8
Description: Extrinsic dental stain area and its intensity were assessed on the facial surfaces of the 6 maxillary and 6 mandibular anterior teeth and the lingual surfaces of the 6 mandibular anterior teeth. Area and intensity of extrinsic dental stain were scored separately for each tooth on the scale 0 to 3, where 0= area with no stain, 1= Stain covering up to one third of area and light intensity stain, 2= Stain covering up to two thirds of area and moderate intensity stain, 3= Stain covering more than two thirds of area and heavy intensity stain. Thus, MLSI score for both Area and Intensity ranged from 0 to 3, where lower score indicated improvement. Change from Baseline was calculated by subtracting the Baseline value from the value at indicated timepoints.
Time Frame: Baseline, Week 4 and Week 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
Number analyzed (Participants) | 92 | 91 | 90
score on a scale
  Area, Week 4 | -0.98 (0.028) | -0.96 (0.028) | -0.09 (0.028)
  Area, Week 8: number analyzed (Participants) | 92 | 91 | 89
  Area, Week 8 | -1.24 (0.026) | -1.30 (0.026) | -0.16 (0.026)
  Intensity, Week 4 | -0.96 (0.023) | -0.96 (0.023) | -0.09 (0.023)
  Intensity, Week 8: number analyzed (Participants) | 92 | 91 | 89
  Intensity, Week 8 | -1.16 (0.024) | -1.21 (0.025) | -0.19 (0.025)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Area, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-0.97 to -0.82], Standard Error of Mean 0.039
Statistical Analysis 2: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Area, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-0.95 to -0.79], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Area, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-1.15 to -1.01], Standard Error of Mean 0.037
Statistical Analysis 4: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Area, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.22 to -1.07], Standard Error of Mean 0.037
Statistical Analysis 5: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Intensity, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-0.93 to -0.80], Standard Error of Mean 0.033
Statistical Analysis 6: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Intensity, Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-0.93 to -0.80], Standard Error of Mean 0.033
Statistical Analysis 7: Comparison: Experimental Dentifrice 1 vs Reference Dentifrice; Intensity, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.04 to -0.90], Standard Error of Mean 0.035
Statistical Analysis 8: Comparison: Experimental Dentifrice 2 vs Reference Dentifrice; Intensity, Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.08 to -0.95], Standard Error of Mean 0.035

ADVERSE EVENTS:
Time Frame: From screening (visit 1) until 5 days following last administration of the study product or last procedure (for approximately 64 days).
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study product including any washout or lead-in product (or medical device).
Groups:
- Experimental Dentifrice 1: Randomized participants were instructed to brush their teeth with the experimental dentifrice 1 (5 % KNO3 dentifrice with 1% alumina and 5% STP), twice daily (morning and evening) for 2 minutes for 8 weeks.
Arm/Group | Experimental Dentifrice 1 | Experimental Dentifrice 2 | Reference Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/92 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/92 | 0/94
Other Adverse Events (participants affected / at risk) | 6/93 | 8/92 | 2/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Dentifrice 1 (N=93) | Experimental Dentifrice 2 (N=92) | Reference Dentifrice (N=94)
ANGULAR CHEILITIS (Gastrointestinal disorders) | 0 | 1 | 0
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 1 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
GINGIVAL SWELLING (Gastrointestinal disorders) | 1 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 1 | 0
LIP EXFOLIATION (Gastrointestinal disorders) | 0 | 1 | 0
LIP PAIN (Gastrointestinal disorders) | 0 | 1 | 0
LIP ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05459558/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT05459558/SAP_001.pdf